CLINICAL TRIAL: NCT04358458
Title: Safety and Efficacy of GEN3009 (DuoHexaBody®-CD37) in Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma - A First-in-Human, Open-label, Phase 1/2a Dose Escalation Trial With Dose Expansion Cohorts
Brief Title: First-in-Human (FIH) Trial of GEN3009 in Subjects With Relapsed or Refractory B-Cell Non-Hodgkin Lymphomas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to strategic evaluation of GEN3009 within context of Genmab's portfolio, decision not based on any safety or regulatory concerns.
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT3009-01; 2019-002752-16 (EudraCT Number); NL72025.056.20 (Registry Identifier: The Netherlands CCMO)
Record Dates: First submitted 2020-04-01; First posted 2020-04-24 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B-cell Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; Small Lymphocytic Lymphoma; Mantle Cell Lymphoma; Chronic Lymphocytic Leukemia; High-grade B-cell Lymphoma; Primary Mediastinal Large B-cell Lymphoma
Keywords: Anti-CD37, monoclonal antibodies, DuoHexabody®
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy Arm (Experimental)
  Interventions: Biological: GEN3009
- Combination Arm (Experimental)
  Interventions: Biological: GEN3009; Biological: Epcoritamab

INTERVENTIONS:
Biological: GEN3009 — GEN3009 will be administered by intravenous (IV) infusion in cycles of 28 days
  Other Names: DuoHexaBody®-CD37
Biological: Epcoritamab — Epcoritamab will be administered by subcutaneous (SC) injections in cycles of 28 days
  Other Names: DuoBody®-CD3xCD20; GEN3013; EPKINLY™
  Arms: Combination Arm

SUMMARY:
The drug that will be investigated in the study is an antibody, GEN3009. Since this is the first study of GEN3009 in humans, the main purpose is to evaluate safety. Besides safety, the study will determine the recommended GEN3009 dose to be tested in a larger group of patients and assess preliminary clinical activity of GEN3009. GEN3009 will be studied in a broad group of cancer patients, having different kinds of lymphomas. All patients will get GEN3009 either as a single treatment (monotherapy) or in combination with another antibody-candidate for treatment of cancer in the blood. The study consists of two parts: Part 1 tests increasing doses of GEN3009 ("escalation"), followed by Part 2 which tests the recommended GEN3009 dose from Part 1 ("expansion").

DETAILED DESCRIPTION:
This trial will be conducted in 2 parts: Part 1 (Dose Escalation) and Part 2 (Dose Expansion). All subjects in Part 1 will receive GEN3009, administered at various dose levels in 28-day cycles. Dose Limiting Toxicity (DLT) will be assessed during the first treatment cycle of Part 1 and the Maximum Tolerated Dose (MTD) and/or Recommended phase 2 dose (RP2D) will be identified.

Subjects in Part 2 will be treated with the Part 1-defined RP2D of GEN3009. Some subjects will receive GEN3009 in combination of a fixed dose of another antibody-candidate. Subjects in Part 2 are assigned either to one of 3 groups: Part 2 Monotherapy (hereafter referred to as 'Part 2A'), Part 2 Combination Safety Run-in ('Part2B') or Part 2 Combination ('Part2C').

Various types of B-cell NHLs are studied, including diffuse large B cell lymphoma (DLBCL), high-grade B cell lymphoma (HGBCL), mantle cell lymphoma (MCL), primary mediastinal large B-cell lymphoma (PMBCL), follicular lymphoma (FL), marginal zone lymphoma (MZL) and chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL).

ELIGIBILITY:
Key Inclusion Criteria:

1. Be at least 18 years of age.
2. Must sign an informed consent form prior to any screening procedures.
3. Dose Escalation: Has histologically or cytologically confirmed relapsed and/or refractory B-cell NHL with no available standard therapy or is not a candidate for available standard therapy, and for whom, in the opinion of the investigator, the experimental therapy may be beneficial. All subjects must have received at least two prior lines of systemic therapy.

   Dose Expansion: Has histologically or cytologically confirmed relapsed or refractory B-cell NHL. All subjects must have received at least 2 prior lines of systemic therapy, and,
   1. For FL and DLBCL, at least 1 of the 2 prior lines of treatment must have been a CD20 containing systemic regimen;
   2. For CLL, subjects must have received at least one prior line of BTK inhibitor or BCL 2 inhibitor.
4. Has one of the eligible subtypes of B-cell NHL :

   Dose Escalation: (DLBCL, HGBCL, PMBCL, FL, MCL, MZL, SLL, or CLL). Dose Expansion: (DLBCL, FL, CLL)
5. Has measurable disease for B-cell NHL or has active disease for Chronic Lymphocytic Leukemia (CLL).
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
7. Has adequate hepatic, renal, and bone marrow functions.
8. Before the first dose of GEN3009, during the trial, and for 12 months after the last dose of GEN3009 and/or the combination, a woman must be either not of childbearing potential or of childbearing potential and practicing a highly effective method of birth control, and must have a negative serum beta-human chorionic gonadotropin (beta-hCG) and urine pregnancy test at screening.
9. A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control.
10. Subjects must have a life expectancy of at least 3 months.

Key Exclusion Criteria:

1. Prior treatment with a CD37-targeting agent.
2. Prior allogeneic Hematopoietic Stem Cell Transplantation (HSCT).
3. Prior treatment with a CD3xCD20 bispecific antibody (Combination Expansion cohort only).
4. Autologous HSCT within 3 months before the first dose of GEN3009.
5. Lymphomas leukemic phase: high absolute lymphocyte count or the presence of abnormal cells in the peripheral blood indicating circulating lymphoma cells.
6. Treatment with an anti-cancer biologic including anti-CD20 therapy, radio-conjugated or toxin-conjugated antibody or chimeric antigen receptor (CAR) T-cell therapy within 4 weeks or 5 half-lives, whichever is shorter, before the first dose of GEN3009. Treatment with small molecules such as BTK inhibitors, BCL2 inhibitors, or PI3K inhibitors within 5 half-lives prior to the first dose of GEN3009.
7. Chemotherapy or radiation therapy within 2 weeks of the first dose of GEN3009.
8. Treatment with an investigational drug or an invasive investigational medical device within 4 weeks or 5 half-lives, whichever is shorter, prior to the first dose of GEN3009, and at any time during the study treatment period.
9. Autoimmune disease or other diseases that require permanent or high-dose immunosuppressive therapy.
10. Received a cumulative dose of corticosteroids more than the equivalent of 250 mg of prednisone within the 2-week period before the first dose of GEN3009.
11. Has uncontrolled intercurrent illness.
12. Seizure disorder requiring therapy (such as steroids or anti-epileptics) (Combination Expansion cohort only).
13. Toxicities from previous anti-cancer therapies have not resolved to baseline levels or to Grade 1 or less except for alopecia and peripheral neuropathy.
14. Primary central nervous system (CNS) lymphoma or known CNS involvement at screening.
15. Known past or current malignancy other than inclusion diagnosis.
16. Had allergic reactions to anti-CD20 or anti-CD37 monoclonal antibody treatment or intolerant to GEN3009 or to the combination therapy excipients.
17. Has had major surgery within 4 weeks before screening or will not have fully recovered from surgery, or has major surgery planned during the time the subject is expected to participate in the trial (or within 4 weeks after the last dose of GEN3009 and/or the combination therapy).
18. Known history/positive serology for hepatitis B.
19. Known medical history or ongoing hepatitis C infection that has not been cured.
20. Known history of seropositivity for HIV infection.
21. Is a woman who is pregnant or breast-feeding, or who is planning to become pregnant while enrolled in this trial or within 12 months after the last dose of GEN3009 and/or the combination therapy.
22. Is a man who plans to father a child while enrolled in this trial or within 12 months after the last dose of GEN3009 and/or the combination therapy.
23. Has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments. Additionally, vulnerable subjects or subjects under guardianship, curatorship, judicial protection or deprived of liberty), are excluded from participation in this trial.
24. Exposed to live/live attenuated vaccine within 4 weeks prior to initiation of GEN3009 treatment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2023-07-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (7):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
- UZ Leuven, Leuven, Belgium
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Odense Universitetshospital, Odense
  - Vejle Sygehus, Vejle
- Amsterdam UMC, Locatie VUMC, Amsterdam, Netherlands
- Spain (5):
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona, L'Hospitalet de Llobregat
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at investigative sites in Belgium, Denmark, France, Spain and the United States from 13 March 2020 to 28 July 2023.
Pre-assignment Details: This study was to be conducted in 2 parts; Part 1 was the dose-escalation phase and Part 2 was the expansion phase. However, the trial was terminated due to strategic evaluation of GEN3009 within context of Genmab's portfolio, the sponsor decided not to conduct the expansion phase (Part 2).
Groups:
- Part 1: GEN3009 Dose Level A in Schedule 1 (S1): Participants received GEN3009 Dose level A in S1 by IV infusion on Days 1, 8, 15, and 22 in cycles 1-3, on Days 1 and 15 in cycles 4-9 and on Day 1 (every 4 weeks) in Cycle 10 until disease progression, unacceptable toxicity, death or end of trial. Each cycle was 28 days in this study.
- Part 1: GEN3009 Dose Level B in S1: Participants received GEN3009 Dose level B in S1 by IV infusion on Days 1, 8, 15, and 22 in cycles 1-3, on Days 1 and 15 in cycles 4-9 and on Day 1 (every 4 weeks) in Cycle 10 until disease progression, unacceptable toxicity, death or end of trial. Each cycle was 28 days in this study.
- Part 1: GEN3009 Dose Level C in S1: Participants received GEN3009 Dose level C in S1 by IV infusion on Days 1, 8, 15, and 22 in cycles 1-3, on Days 1 and 15 in cycles 4-9 and on Day 1 (every 4 weeks) in Cycle 10 until disease progression, unacceptable toxicity, death or end of trial. Each cycle was 28 days in this study.
- Part 1: GEN3009 Dose Level D in S1: Participants received GEN3009 Dose level D in S1 by IV infusion on Days 1, 8, 15, and 22 in cycles 1-3, on Days 1 and 15 in cycles 4-9 and on Day 1 (every 4 weeks) in Cycle 10 until disease progression, unacceptable toxicity, death or end of trial. Each cycle was 28 days in this study. For cycle 1, participants received the dose split into 2 consecutive days. i.e., at Cycle 1 Day 1 (C1D1) and the remaining amount at Day 2 (C1D2).
- Part 1: GEN3009 Dose Level D in Schedule (S2): Participants received GEN3009 Dose level D in S2 (in US only) by IV infusion on Days 1, 4, 8, 11, 15, 18, 22 and 25 in cycles 1, Day 1, 8, 15 and 22 in Cycles 2-3, Day 1 and 15 in Cycles 4-9 and Day 1 starting Cycle 10 until disease progression, unacceptable toxicity, death or end of trial. Each cycle was 28 days in this study. Participants received half of the full dose on Days 1, 4, 8, 11, 15, 18, 22, and 25 i.e. two half doses on Days 1 and 4 of each week for the first cycle.
- Part 1: GEN3009 Dose Level E in S1: Participants received GEN3009 Dose level E in S1 by IV infusion on Days 1, 8, 15, and 22 in cycles 1-3, on Days 1 and 15 in cycles 4-9 and on Day 1 (every 4 weeks) in Cycle 10 until disease progression, unacceptable toxicity, death or end of trial. Each cycle was 28 days in this study. For cycle 1, participants received the dose split into 2 consecutive days. i.e., at C1D1 and the remaining amount at C1D2.
- Part 1: GEN3009 Dose Level F in S1: Participants received GEN3009 Dose level F in S1 by IV infusion on Days 1, 8, 15, and 22 in cycles 1-3, on Days 1 and 15 in cycles 4-9 and on Day 1 (every 4 weeks) in Cycle 10 until disease progression, unacceptable toxicity, death or end of trial. Each cycle was 28 days in this study. For cycle 1, participants received the dose split into 2 consecutive days. i.e., at C1D1 and the remaining amount at C1D2.
- Part 1: GEN3009 Dose Level G in S1: Participants received GEN3009 Dose level G in S1 by IV infusion on Days 1, 8, 15, and 22 in cycles 1-3, on Days 1 and 15 in cycles 4-9 and on Day 1 (every 4 weeks) in Cycle 10 until disease progression, unacceptable toxicity, death or end of trial. Each cycle was 28 days in this study. For cycle 1, participants received the dose split into 2 consecutive days. i.e., at C1D1 and the remaining amount at C1D2.
Period: Overall Study
Arm/Group | Part 1: GEN3009 Dose Level A in Schedule 1 (S1) | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in Schedule (S2) | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Started | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
Not completed — Death | 1 | 1 | 3 | 8 | 1 | 6 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Site is closing study participation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor request | 2 | 3 | 3 | 0 | 2 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) comprises all participants to whom study drug had been assigned and who had received at least 1 dose of GEN3009.
Groups:
- Part 1: GEN3009 Dose Level A in S1: Participants received GEN3009 Dose level A in S1 by IV infusion on Days 1, 8, 15, and 22 in cycles 1-3, on Days 1 and 15 in cycles 4-9 and on Day 1 (every 4 weeks) in Cycle 10 until disease progression, unacceptable toxicity, death or end of trial. Each cycle was 28 days in this study.
- Part 1: GEN3009 Dose Level D in S1: Participants received GEN3009 Dose level D in S1 by IV infusion on Days 1, 8, 15, and 22 in cycles 1-3, on Days 1 and 15 in cycles 4-9 and on Day 1 (every 4 weeks) in Cycle 10 until disease progression, unacceptable toxicity, death or end of trial. Each cycle was 28 days in this study. For cycle 1, participants received the dose split into 2 consecutive days. i.e., at C1D1 and the remaining amount at C1D2.
- Part 1: GEN3009 Dose Level D in S2: Participants received GEN3009 Dose level D in S2 (in US only) by IV infusion on Days 1, 4, 8, 11, 15, 18, 22 and 25 in cycles 1, Day 1, 8, 15 and 22 in Cycles 2-3, Day 1 and 15 in Cycles 4-9 and Day 1 starting Cycle 10 until disease progression, unacceptable toxicity, death or end of trial. Each cycle was 28 days in this study. Participants received half of the full dose on Days 1, 4, 8, 11, 15, 18, 22, and 25 i.e. two half doses on Days 1 and 4 of each week for the first cycle.
- Total: Total of all reporting groups
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1 | Total
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (3.46) | 54.5 (8.81) | 74.6 (8.68) | 67.1 (9.89) | 63.3 (16.86) | 69.4 (10.23) | 70.3 (9.87) | 60.8 (17.38) | 66.7 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 2 | 0 | 2 | 1 | 1 | 11
  Male | 1 | 3 | 5 | 8 | 3 | 8 | 2 | 5 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Missing | 0 | 2 | 5 | 4 | 0 | 8 | 3 | 3 | 25
  Ethnicity: Not Hispanic or Latino | 2 | 2 | 2 | 6 | 3 | 0 | 0 | 3 | 18
  Ethnicity: Not Reported | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 5
  Race: Missing | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Race: Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Race: Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Race: White | 2 | 3 | 7 | 7 | 3 | 8 | 3 | 5 | 38
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Denmark | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 1 | 7
  Netherlands | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 6
  Spain | 0 | 2 | 3 | 1 | 0 | 3 | 1 | 0 | 10
  United States | 3 | 2 | 2 | 6 | 3 | 2 | 0 | 3 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs were graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, except for TLS (Cairo-Bishop grading) and CRS/ICANS (Lee et al., 2019). These criteria include: all Grade 5 toxicities; hematologic events including thrombocytopenia Grade 4, neutropenia Grade 4, Febrile neutropenia Grade 3 or 4, Grade 3 or 4 hemorrhage associated with thrombocytopenia of ≥Grade 3, anemia of Grade 4 and tumor lysis syndrome (TLS) Grade 4; and non-hematologic AEs of Grade 3 or higher excluding certain fevers, hypotension, laboratory values, Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT), nausea, vomiting, diarrhea, fatigue/asthenia, or alopecia (no grading), which meet certain additional criteria.
Time Frame: During the first treatment cycle (Cycle length=28 days)
Population: The Safety analysis set included all participants who had received at least 1 dose of GEN3009.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE is any untoward medical occurrence in a clinical trial participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as an AE that meets one of the following criteria: is fatal or life-threatening; results in persistent or significant disability/incapacity; constitutes a congenital anomaly/birth defect; is medically significant (an event that jeopardizes the participant or may require medical or surgical intervention to prevent one of the outcomes listed above [medical and scientific judgment must be exercised in deciding whether an AE is "medically significant"]); required inpatient hospitalization or prolongation of existing hospitalization. TEAEs are defined as AEs which begin, or worsen, during the on-treatment period ending 4 weeks after the last dose of study medication.
Time Frame: From first dose until 30 days after the last dose (up to 15.5 months)
Population: The Safety analysis set included all participants who had received at least 1 dose of GEN3009.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
Participants
  Participants with TEAEs | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
  Participants with Serious TEAEs | 0 | 0 | 4 | 7 | 2 | 4 | 2 | 4

3. Primary Outcome: Number of Participants With AEs of Special Interest (AESI)
Description: AESIs are defined as events (serious or non-serious) that are of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor may be appropriate.
Time Frame: From first dose until 30 days after the last dose (up to 15.5 months)
Population: The Safety analysis set included all participants who had received at least 1 dose of GEN3009.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
Participants | 1 | 1 | 7 | 9 | 3 | 10 | 3 | 5

4. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities Reported as TEAEs
Description: Laboratory parameters included hematology, serum chemistries and urinalysis. Clinically significant laboratory abnormalities were based upon the Investigator's discretion. Laboratory parameters captured as AEs are reported in this outcome measure.
Time Frame: From first dose until 30 days after the last dose (up to 15.5 months)
Population: The Safety analysis set included all participants who had received at least 1 dose of GEN3009.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
Participants
  Blood creatinine increased | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
  Blood alkaline phosphatase increased | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  Blood lactate dehydrogenase increased | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Alanine aminotransferase increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood creatine increased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

5. Primary Outcome: Number of Participants With Clinically Notable Vital Signs
Description: Criteria for clinically notable (elevated and below normal values respectively) vital signs are as follows: Systolic Blood Pressure (SBP): ≥180 millimeters of mercury (mmHg) and an increase ≥20 mmHg from baseline, ≤90 mmHg and a decrease ≥20 mmHg from baseline; Diastolic Blood Pressure (DBP): ≥105 mmHg and an increase ≥15 mmHg from baseline, ≤50 mmHg and a decrease ≥15 mmHg from baseline; Heart rate: ≥120 beats per minute (bpm) with an increase of ≥15 bpm from baseline, ≤50 bpm and a decrease ≥15 bpm from baseline; Temperature: > 38 degree Celsius (°C) and < 35°C. Number of participants with clinically notable elevated and below normal vital signs values up to end of treatment are reported.
Time Frame: From first dose up to end of treatment (up to 14.5 months)
Population: The Safety analysis set included all participants who had received at least 1 dose of GEN3009. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 5 | 9 | 3 | 8 | 2 | 5
Participants
  SBP: Elevated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP: Below Normal | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1
  DBP: Elevated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP: Below Normal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Heart Rate: Elevated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Heart Rate: Below Normal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Elevated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Below Normal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Dose Delays and Dose Interruptions
Description: Number of participants with dose delays and dose Interruptions due to AE, Coronavirus disease 2019 (COVID-19), drug administration issues and other unspecified reasons are reported.
Time Frame: From first dose until 30 days after the last dose (up to 15.5 months)
Population: The Safety analysis set included all participants who had received at least 1 dose of GEN3009.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
Participants
  Dose delay due to AE | 0 | 0 | 4 | 1 | 1 | 2 | 1 | 2
  Dose delay due to Coronavirus disease 2019 (COVID-19) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dose delay due to un-specified reason | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
  Dose interruption due to AE | 0 | 1 | 7 | 9 | 3 | 10 | 3 | 5
  Dose interruption due to drug administration issues | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Dose interruption due to unspecified reason | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

7. Primary Outcome: Actual Dose Intensity
Description: Actual dose intensity (milligrams per cycle [mg/cycle]) is calculated as cumulative dose/number of cycles initiated.
Time Frame: From first dose until 30 days after the last dose (up to 15.5 months)
Population: The Safety analysis set included all participants who had received at least 1 dose of GEN3009. 'Number analyzed' indicates the number of participants with data available for analysis at specified cycle duration.
Measure: Mean (Standard Deviation); unit: mg/cycle
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
mg/cycle
  Cycles 1-3 | 114.67 (112.10) | 720.00 (0.00) | 1389.46 (278.91) | 2501.53 (992.91) | 2515.85 (1053.90) | 3903.62 (1135.72) | 5957.23 (766.90) | 6973.78 (1072.58)
  Cycles 4-9: number analyzed (Participants) | 0 | 1 | 4 | 1 | 0 | 1 | 2 | 0
  Cycles 4-9 |  | 363.71 (NA) — Since there is only 1 participant, standard deviation (SD) was not estimable. | 799.71 (10.64) | 1527.27 (NA) — Since there is only 1 participant, SD was not estimable. |  | 2400.00 (NA) — Since there is only 1 participant, SD was not estimable. | 2953.02 (349.28) |
  Cycle 10-until end of study: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 10-until end of study |  |  | 318.94 (NA) — Since there is only 1 participant, SD was not estimable. |  |  |  |  |

8. Secondary Outcome: Apparent Total Plasma Clearance (CL) of GEN3009
Time Frame: Pre-dose and 5 minutes post-dose on days 1, 2, 4 (S2 only), 8, 15, 22 and 2 hours (h) and 4h post-dose on days 1 and 2, 24h post-dose on day 2 and 72h post-dose on day 4 of Cycles 1 and 2 (Each cycle length=28 days)
Population: The pharmacokinetic analysis set (PAS) includes all participants who have been exposed to GEN3009 and have had at least one pharmacokinetic sample collected that has provided a valid bioanalytical result.
Measure: Mean (Standard Deviation); unit: Liters per day
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
Liters per day
  Cycle 1 | NA (NA) — Data was not estimable because the values were below the lower limit of quantification (LLOQ). | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ.
  Cycle 2 | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ.

9. Secondary Outcome: Volume of Distribution of GEN3009
Time Frame: Pre-dose and 5 minutes post-dose on days 1, 2, 4 (S2 only), 8, 15, 22 and 2h and 4h post-dose on days 1 and 2, 24h post-dose on day 2 and 72h post-dose on day 4 of Cycles 1 and 2 (Each cycle length=28 days)
Population: The PAS includes all participants who have been exposed to GEN3009 and have had at least one pharmacokinetic sample collected that has provided a valid bioanalytical result.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
mL
  Cycle 1 | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ.
  Cycle 2 | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ.

10. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Day 7 of GEN3009
Time Frame: Pre-dose and 5 minutes post-dose on days 1, 2 and 4 (S2 only); 2h and 4h post-dose on days 1 and 2, 24h post-dose on day 2 and 72h post-dose on day 4 of Cycles 1 and 2 (Each cycle length=28 days)
Population: The PAS includes all participants who have been exposed to GEN3009 and have had at least one pharmacokinetic sample collected that has provided a valid bioanalytical result. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants with data available for analysis at a specified cycle.
Measure: Mean (Standard Deviation); unit: micrograms*day per milliliter(ug*day/mL)
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 0 | 0 | 3 | 2 | 1 | 2 | 3 | 3
micrograms*day per milliliter(ug*day/mL)
  Cycle 1: number analyzed (Participants) | 0 | 0 | 2 | 1 | 1 | 2 | 3 | 3
  Cycle 1 |  |  | 159.2796 (95.7330) | 181.5966 (NA) — Since there is only 1 participant, SD was not estimable. | 260.8704 (NA) — Since there is only 1 participant, SD was not estimable. | 219.1863 (46.3749) | 353.5017 (177.2169) | 389.0321 (126.8407)
  Cycle 2: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 2 | 3 | 0
  Cycle 2 |  |  | 132.6580 (NA) — Since there is only 1 participant, SD was not estimable. | 159.3302 (22.1333) |  | 159.3456 (98.0641) | 363.4413 (190.0120) |

11. Secondary Outcome: AUC From Time 0 to Infinity (AUCinf) of GEN3009
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ug*day/mL
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 2 | 4 | 7 | 8 | 3 | 8 | 3 | 5
ug*day/mL
  Cycle 1: number analyzed (Participants) | 2 | 4 | 6 | 7 | 2 | 7 | 3 | 5
  Cycle 1 | 6.0154 (3.8503) | 56.3289 (22.4400) | 136.8615 (72.7498) | 163.9206 (52.0135) | 332.1408 (73.1435) | 192.0412 (90.3476) | 358.0010 (183.3857) | 335.8745 (117.1831)
  Cycle 2: number analyzed (Participants) | 2 | 3 | 5 | 4 | 3 | 5 | 3 | 0
  Cycle 2 | 5.9939 (0.6498) | 46.4191 (9.8966) | 139.9286 (61.7235) | 127.4566 (49.8017) | 957.4149 (1427.7939) | 159.8668 (73.6559) | 363.7766 (190.3613) |

12. Secondary Outcome: AUC From Time 0 to Time of Last Dose (AUClast) of GEN3009
Time Frame: as for outcome 9
Population: The PAS includes all participants who have been exposed to GEN3009 and have had at least one pharmacokinetic sample collected that has provided a valid bioanalytical result. 'Number analyzed' indicates the number of participants with data available for analysis at specified cycle duration.
Measure: Mean (Standard Deviation); unit: ug*day/mL
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
ug*day/mL
  Cycle 1: number analyzed (Participants) | 2 | 4 | 7 | 8 | 3 | 9 | 3 | 6
  Cycle 1 | 4.5524 (2.3467) | 51.0701 (17.1901) | 103.4129 (73.3627) | 148.4079 (41.7750) | 467.9622 (283.7778) | 150.7393 (96.0893) | 353.5017 (177.2169) | 327.1762 (109.9472)
  Cycle 2: number analyzed (Participants) | 2 | 3 | 5 | 5 | 3 | 5 | 3 | 0
  Cycle 2 | 4.4707 (1.3098) | 45.0924 (9.1404) | 121.5349 (53.0658) | 103.5413 (61.7884) | 441.7798 (542.0539) | 152.4631 (74.1040) | 363.4413 (190.0120) |

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of GEN3009
Time Frame: as for outcome 9
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: microgram per milliliter (ug/mL)
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
microgram per milliliter (ug/mL)
  Cycle 1: number analyzed (Participants) | 2 | 4 | 7 | 8 | 3 | 9 | 3 | 6
  Cycle 1 | 8.3000 (3.5355) | 43.4000 (12.7674) | 89.8714 (39.8257) | 139.0000 (43.8341) | 363.0667 (460.6843) | 144.4778 (79.0905) | 317.3333 (51.4328) | 352.6667 (58.5514)
  Cycle 2: number analyzed (Participants) | 2 | 3 | 5 | 5 | 3 | 5 | 3 | 0
  Cycle 2 | 8.1050 (3.6699) | 46.1667 (2.7934) | 118.4800 (29.9458) | 147.4000 (52.7286) | 572.0000 (708.4659) | 237.0000 (30.8869) | 394.6667 (109.5871) |

14. Secondary Outcome: Time to Reach Cmax (Tmax) of GEN3009
Time Frame: as for outcome 9
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
days
  Cycle 1: number analyzed (Participants) | 2 | 4 | 7 | 8 | 3 | 9 | 3 | 6
  Cycle 1 | 0.0765 (0.0120) | 0.1490 (0.0957) | 0.2084 (0.0553) | 0.6039 (0.6768) | 1.2123 (1.5987) | 0.5030 (0.2908) | 1.3817 (0.0890) | 1.2580 (0.0771)
  Cycle 2: number analyzed (Participants) | 2 | 3 | 5 | 5 | 3 | 5 | 3 | 0
  Cycle 2 | 0.0445 (0.0007) | 0.1650 (0.1643) | 0.1656 (0.0820) | 0.2740 (0.3010) | 0.2030 (0.0346) | 0.1620 (0.0595) | 0.1983 (0.0535) |

15. Secondary Outcome: Trough Concentrations (Ctrough) of GEN3009
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
ug/mL
  Cycle 1 | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ.
  Cycle 2 | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ.

16. Secondary Outcome: Terminal Elimination Half-Life (t 1/2) of GEN3009
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
days
  Cycle 1 | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ.
  Cycle 2 | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ. | NA (NA) — Data was not estimable because the values were below the LLOQ.

17. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADAs)
Description: Venous blood samples will be collected for measurement of serum concentrations of ADAs. Number of participants with positive ADAs are reported in this outcome measure. The detection of ADAs was performed using validated, specific and sensitive Electrochemiluminescence Immunoassay (ECLIA) method.
Time Frame: From first dose until 30 days after the last dose (up to 15.5 months)
Population: The immunogenicity analysis set included all participants who had received at least 1 dose of study drug and had a baseline and at least 1 evaluable on-treatment ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 3 | 7 | 8 | 3 | 9 | 3 | 3
Participants | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0

18. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time from the first documentation of objective tumor response [Complete response (CR) or Partial response (PR)] to the date of first disease progression (PD) or death as assessed by the investigator based on Lugano criteria for B-cell non-Hodgkin lymphoma (B-cell NHL) and International Workshop on Chronic Lymphocytic Leukemia (iwCLL) for chronic lymphocytic leukemia (CLL). Detailed definition of CR, PR and PD as per Lugano and iwCLL criteria in the protocol appendices.
Time Frame: From date of first documented CR or PR up to disease progression or death (up to approximately 3 years 4 months)
Population: The FAS comprises all participants to whom study drug had been assigned and who had received at least 1 dose of GEN3009. 'Overall number of participants Analyzed' signified the participants who achieved CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 0 | 0 | 3 | 0 | 1 | 3 | 2 | 1
months |  |  | 15.9 [2.9 to NA] — Upper limit of confidence interval (CI) not reached due to less number of participants with events. |  | NA [NA to NA] — Median, upper and lower limit of CI not reached due to less number of participants with events. | 1.4 [1.4 to NA] — Upper limit of confidence interval CI not reached due to less number of participants with events. | NA [NA to NA] — Median, upper and lower limit of CI not reached due to less number of participants with events. | 4.1 [NA to NA] — Upper and lower limit of CI not reached due to less number of participants with events.

19. Secondary Outcome: Time to Response (TTR)
Description: TTR: time from first dose of administration until date of first response as assessed by investigator based on Lugano criteria for B-cell NHL and iwCLL for CLL. It is derived for all participants who achieved PR or CR. Detailed definitions of CR, PR and PD as per Lugano and iwCLL criteria in the protocol appendices.
Time Frame: From date of first documented CR or PR up to disease progression or death (up to approximately 3 years 4 months)
Population: The FAS comprises all participants to whom study drug had been assigned and who had received at least 1 dose of GEN3009. 'Overall number of participants analyzed' indicates the number of participants who achieved CR or PR.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 0 | 0 | 3 | 0 | 1 | 3 | 2 | 1
months |  |  | 1.3361 (0.1004) |  | 1.8727 (NA) — Since there is only 1 participant, SD was not estimable. | 1.2704 (0.2138) | 2.0370 (1.0222) | 1.1828 (NA) — Since there is only 1 participant, SD was not estimable.

20. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time in days from Day 1 of Cycle 1 to the day of first documented PD, or the day of death due to any cause, whichever comes first as assessed by investigator based on Lugano Criteria for B-cell NHL and iwCLL for CLL. PFS was estimated using the Kaplan-Meier method. Detailed definitions of PD as per Lugano and iwCLL criteria in the protocol appendices.
Time Frame: From day of first dose until disease progression or death due to any cause (up to approximately 3 years 4 months)
Population: The FAS comprises all participants to whom study drug had been assigned and who had received at least 1 dose of GEN3009.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
months | 1.4 [1.2 to NA] — Upper limit of CI not reached due to less number of participants with events. | 2.6 [1.3 to NA] — Upper limit of CI not reached due to less number of participants with events. | 4.3 [1.8 to NA] — Upper limit of CI not reached due to less number of participants with events. | 1.2 [1.0 to 4.0] | 2.3 [1.4 to NA] — Upper limit of CI not reached due to less number of participants with events. | 1.9 [0.2 to 3.4] | NA [1.3 to NA] — Median and upper limit of CI not reached due to less number of participants with events. | 0.8 [0.4 to NA] — Upper limit of CI not reached due to less number of participants with events.

21. Secondary Outcome: Overall Survival (OS)
Description: The OS is defined as the time from the start of study treatment until death due to any cause. The OS was estimated using Kaplan-Meier method.
Time Frame: From day of first dose until disease progression or death due to any cause (up to approximately 3 years 4 months)
Population: The FAS comprises all participants to whom study drug had been assigned and who had received at least 1 dose of GEN3009.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 4 | 7 | 10 | 3 | 10 | 3 | 6
months | NA [19.1 to NA] — Upper limit of CI not reached due to less number of participants with events. | NA [5.2 to NA] — Median and upper and limit of CI not reached due to less number of participants with events. | NA [1.8 to NA] — Median and upper and limit of CI not reached due to less number of participants with events. | 10.9 [0.8 to 18.0] | NA [14.0 to NA] — Upper limit of CI not reached due to less number of participants with events. | 13.7 [0.2 to NA] — Upper limit of CI not reached due to less number of participants with events. | 13.1 [7.0 to NA] — Upper limit of CI not reached due to less number of participants with events. | 6.6 [0.5 to NA] — Upper limit of CI not reached due to less number of participants with events.

22. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR: the percentage of participants who achieved a best overall response (BOR) of CR or PR as assessed by investigator based on Lugano Criteria for B-cell NHL and iwCLL for CLL. Detailed definitions of CR and PR as per Lugano and iwCLL criteria in the protocol appendices.
Time Frame: From day of first dose until disease progression or death due to any cause (up to approximately 3 years 4 months)
Population: The Response Evaluable Set includes all participants in FAS who have baseline evaluable disease and had at least 1 post-baseline disease evaluation or died within 60 days of first trial treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 3 | 7 | 8 | 3 | 8 | 3 | 6
percentage of participants | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 42.9 [9.9 to 81.6] | 0 [0.0 to 36.9] | 33.3 [0.8 to 90.6] | 37.5 [8.5 to 75.5] | 66.7 [9.4 to 99.2] | 16.7 [0.4 to 64.1]

23. Secondary Outcome: CR Rate
Description: CR rate was estimated using Clopper-Pearson method. Detailed definitions of CR as per Lugano and iwCLL criteria in the protocol appendices.
Time Frame: From day of first dose until disease progression or death due to any cause (up to approximately 3 years 4 months)
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
Number analyzed (Participants) | 3 | 3 | 7 | 8 | 3 | 8 | 3 | 6
percentage of participants | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 28.6 [3.7 to 71.0] | 0 [0.0 to 36.9] | 33.3 [0.8 to 90.6] | 0 [0.0 to 36.9] | 33.3 [0.8 to 90.6] | 0 [0.0 to 45.9]

ADVERSE EVENTS:
Time Frame: Deaths were assessed up to approximately 3 years, 4 months; Adverse Events were assessed up to 15.5 months
Description: The Safety analysis set included all participants who had received at least 1 dose of GEN3009.
Groups:
- Part 1: GEN3009 Dose Level E in S1: Participants received GEN3009 Dose level E in S1 by IV infusion on Days 1, 8, 15, and 22 in cycles 1-3, on Days 1 and 15 in cycles 4-9 and on Day 1 (every 4 weeks) in Cycle 10 until disease progression, unacceptable toxicity, death or end of trial. Each cycle was 8 days in this study. For cycle 1, participants received the dose split into 2 consecutive days. i.e., at C1D1 and the remaining amount at C1D2.
Arm/Group | Part 1: GEN3009 Dose Level A in S1 | Part 1: GEN3009 Dose Level B in S1 | Part 1: GEN3009 Dose Level C in S1 | Part 1: GEN3009 Dose Level D in S1 | Part 1: GEN3009 Dose Level D in S2 | Part 1: GEN3009 Dose Level E in S1 | Part 1: GEN3009 Dose Level F in S1 | Part 1: GEN3009 Dose Level G in S1
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/4 | 3/7 | 8/10 | 1/3 | 6/10 | 2/3 | 3/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 4/7 | 7/10 | 2/3 | 4/10 | 2/3 | 4/6
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 7/7 | 9/10 | 3/3 | 10/10 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: GEN3009 Dose Level A in S1 (N=3) | Part 1: GEN3009 Dose Level B in S1 (N=4) | Part 1: GEN3009 Dose Level C in S1 (N=7) | Part 1: GEN3009 Dose Level D in S1 (N=10) | Part 1: GEN3009 Dose Level D in S2 (N=3) | Part 1: GEN3009 Dose Level E in S1 (N=10) | Part 1: GEN3009 Dose Level F in S1 (N=3) | Part 1: GEN3009 Dose Level G in S1 (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: GEN3009 Dose Level A in S1 (N=3) | Part 1: GEN3009 Dose Level B in S1 (N=4) | Part 1: GEN3009 Dose Level C in S1 (N=7) | Part 1: GEN3009 Dose Level D in S1 (N=10) | Part 1: GEN3009 Dose Level D in S2 (N=3) | Part 1: GEN3009 Dose Level E in S1 (N=10) | Part 1: GEN3009 Dose Level F in S1 (N=3) | Part 1: GEN3009 Dose Level G in S1 (N=6)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scleral haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Refractive amblyopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Injection site phlebitis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 2 | 3 | 0 | 3 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 7 | 9 | 3 | 7 | 3 | 6
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meralgia paraesthetica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 4 | 0 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Feeling jittery (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vein disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 3 | 1 | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 7 | 7 | 3 | 10 | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 3 | 0 | 4 | 0 | 2
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion site paraesthesia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 3 | 6 | 0 | 6 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The trial was terminated due to strategic evaluation of GEN3009 within context of Genmab's portfolio, decision not based on any safety or regulatory concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT04358458/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT04358458/SAP_001.pdf